CLINICAL TRIAL: NCT05899504
Title: The Use of Novel Over-The-Scope-Clip to Prevent Esophageal Stent Migration- Randomized Controlled Trial- A Pilot Study
Brief Title: The Use of Novel Over-The-Scope-Clip to Prevent Esophageal Stent Migration
Acronym: NOTSC-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Collaborators: Ovesco Endoscopy AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NOTSC-01
Record Dates: First submitted 2023-01-29; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Migration of Implant

STUDY DESIGN:
Intervention Model Description: A new endoscopic clipping device called the over-the-scope-clip (OTSC) system (Ovesco Endoscopy, Tübingen, Germany) has become available for the closure of perforations, anastomotic leaks, and fistulas. The OTSC system has a stronger closing force than the through-the-scope hemostatic clip. Therefore, some researchers have reported esophageal SEMS fixation with an OTSC to prevent migration
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Interventional) Patients undergoing Esophageal stenting with over the scope clip (OTSC) stent fix (Experimental): Marking clips will be placed with endoscopy at the upper end of the stricture. In mild stricture cases that allowed the passage of the endoscope, marking clips will also placed in the lower end. A stent that of at least 4 cm longer than the stricture will be used to allow at least a 2-cm extension above and below the proximal and distal tumor margins. The stent positioned over a guidewire and deployed under fluoroscopy guidance and, in some cases, also under endoscopy guidance. Subsequently, the OTSC system will be loaded onto the scope and part of the upper rim of the stent will be suctioned into the transparent cap before releasing the OTSC, grasping both the SEMS and esophageal wall. Investigator will avoid deploying the OTSC in areas of pulsations to prevent potential grasping of the vasculature structure. Only a single OTSC will be placed per participants.
  Interventions: Device: Over-The-Scope-Clip (OTSC) Stent Fix
- (Non- Interventional) Participants undergoing Esophageal stenting without OTSC stent fix (No Intervention): This will be the standard procedure of esophageal stent placement under fluro imaging/screening

INTERVENTIONS:
Device: Over-The-Scope-Clip (OTSC) Stent Fix — A stent that of at least 4 cm longer than the stricture will be used to allow at least a 2-cm extension above and below the proximal and distal tumor margins. The stent positioned over a guidewire and deployed under fluoroscopy guidance and, in some cases, also under endoscopy guidance. Subsequently, the OTSC system will be loaded onto the scope and part of the upper rim of the stent will be suctioned into the transparent cap before releasing the OTSC, grasping both the SEMS and esophageal wall. We will avoid deploying the OTSC in areas of pulsations to prevent potential grasping of the vasculature structure
  Arms: (Interventional) Patients undergoing Esophageal stenting with over the scope clip (OTSC) stent fix

SUMMARY:
New endoscopic clipping device called the over-the-scope-clip (OTSC) system (Ovesco Endoscopy, Tübingen, Germany) has become available for the closure of perforations, anastomotic leaks, and fistulas. The OTSC system has a stronger closing force than the through-the-scope hemostatic clip. Therefore, some researchers have reported esophageal SEMS fixation with an OTSC to prevent migration.

DETAILED DESCRIPTION:
Participants requiring esophageal SEMS placement for various indications such as stricture (benign, malignant), leaks All participants who require esophageal SEMS placement. Esophago-gastroscopy will be done to assess the feasibility of SEMS placement.

Participants are randomized into two arms- one arm (interventional) use of OTSC stent fix after esophageal SEMS placement or the other arm (non-interventional) esophageal SEMS is placed.

Participants are followed up for 1 year to observe stent migration rate in both the groups.

ELIGIBILITY:
Inclusion Criteria:

* All adults (18+ years)
* Have benign, malignant non-stricture esophageal lesions (i.e. fistulae, perforation, leaks) warranting esophageal stent placement as an inpatient or outpatient
* Ability to consent to stent fixation.

Exclusion Criteria:

* Patients aged under 18 years of age
* Unable to provide informed consent
* Inherited or acquired coagulopathy likely to affect the risk of bleeding
* Receiving anticoagulant therapy that could not be stopped or bridged prior to procedure
* Breast feeding, pregnant and lactating women's.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Esophageal SEMS migration rate at 4 weeks follow up. | 4 weeks
  Proportion of patients experiencing stent migration at 4 weeks after index procedure.

SECONDARY OUTCOMES:
Procedural time in minutes | immediately after procedure
  Total time required to complete the intended procedure
Migration of stent in both groups | 6 months
  Time to migration after stent placement in respective groups
Adverse events in both groups apart from stent migration | 6 months
  All the adverse events will be recorded, excluding SEMS migration, which is already an primary outcome measure separately
Improvement in dysphagia score | 1 week
  Improvement in dysphagia score at one week post procedure in both the arms